CLINICAL TRIAL: NCT02200744
Title: Incidence of Recall After Procedural Sedation With Propofol in the Emergency Department
Acronym: MEMOPROPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/CHU/08; 2013-003669-32 (Other: Agence National de Sécurité du Médicament)
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Fractures Reduction; Joint Dislocation Reduction
Keywords: Procedural sedation; emergency department; adults; propofol; recall assessment
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dislocation reduction using propofol

SUMMARY:
The purpose of this study is to determine the incidence of recall in patients managed in emergency department with a procedural sedation protocol using propofol in a population of 250 .

DETAILED DESCRIPTION:
After procedural sedation for fracture or joint dislocation reduction using propofol, adult patients recall will be assessed with a standardised form. This recall assessment will be realised 2 hours (+/- 15 minutes) after the procedural sedation and the day after.

The primary outcome measure will be the recall incidence 2 hours (+/- 15 minutes) after a procedural sedation. A secondary outcome will be the recall incidence one day after the procedural sedation.

The recall will be defined by a positive answer to the third question of the Sandin form (Lancet. 2000;355(9205):707-11).

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (> 18 years old) who had a procedural sedation in emergency department using propofol for fracture or joint dislocation reduction
* Patients who received an initial injection of Propofol by slow intravenous injection of 1 mg/kg in 20 seconds
* Inclusion less than 2 hours from the injection of Propofol
* Patients who have signed a consent to participate in the study
* Patients covered by social security.

Exclusion Criteria:

* Patients under 18 years old
* Patients who cannot signed the informed consent
* Patients who had procedural sedation using other drugs that propofol
* Participation in another study type biomedical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients managed in emergency department with a procedural sedation protocol using propofol
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Recall incidence | At 2 hours (+/- 15 minutes) after procedural sedation with propofol
  questionnaire of Brice amended by Sandin

SECONDARY OUTCOMES:
Recall incidence | About 24 hours after procedural sedation with propofol
  The patient will be contacted by phone the next day after procedural sedation with propofol. They will answer the questionnaire of Brice amended by Sandin
Patient's satisfaction assessment | At 2 hours (+/- 15 minutes) after procedural sedation with propofol
  numerical verbal scale

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Jean Marianne, MD, Principal Investigator — CHU de La Réunion; Marc Weber, MD, Principal Investigator — Groupe Hospitalier Est Réunion; Katia Mougin, MD, Principal Investigator — Centre Hospitalier Gabriel Martin
Locations (4):
- France (4):
  - Groupe Hospitalier Est Réunion, Saint-Benoît, La Réunion
  - CHU de la Réunion, Saint-Denis, La Réunion
  - Centre Hospitalier Gabriel Martin, Saint-Paul, La Réunion
  - CHU de La Réunion, Saint-Pierre, La Réunion

REFERENCES:
- [Derived] Muller B, Mougin K, Weber M, Beti E, Guihard B, Tounkara BS, Combes X. Recall Incidence After Procedural Sedation With Propofol in Emergency Departments. J Emerg Med. 2025 Dec;79:457-462. doi: 10.1016/j.jemermed.2025.09.013. Epub 2025 Sep 9. PMID 41205307